CLINICAL TRIAL: NCT02628821
Title: Effectiveness of Synchronized Non-Invasive Ventilation to Prevent Invasive Mechanical Ventilation Use in Preterm Infants.
Brief Title: The Effectiveness of Non-Invasive Ventilation Use in Preterm Infants.
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Manuel Sanchez Luna, Dr., Hospital General Universitario Gregorio Marañon
Other Study IDs: 02/2015
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Noninvasive Ventilation; Preterm Infants
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preterm Infants treated with non-invasive ventilation: Preterm Infants of less than 32 weeks of Gestational age treated with synchronized non-invasive ventilation (SNIPPV) to prevent intubation or extubation failure based in a prospective protocol:
  * nCPAP failure: Preterm infants supported with nCPAP that meet intubation criteria if they are in a stable situation.
  * Electively For extubation:
  Preterm infants in which nCPAP extubation has previously failed or Prolonged mechanical ventilation (more than 15 days) with high respiratory parameters (PMAP > 10 cmH2O and FiO2>35%).
  Interventions: Other: Preterm Infants treated with non-invasive ventilation.

INTERVENTIONS:
Other: Preterm Infants treated with non-invasive ventilation.
  Other Names: (Giulia®, Neonatal Nasal Ventilator)

SUMMARY:
Prospective observational study of SNIPPV use in preterm infants of less than 32weeks of gestation from January 2012 to December 2015. Previous respiratory status is analyzed as well as respiratory outcomes and possible secondary side effects.

SNIPPV is used to prevent Intubation in Infants in which nCPAP has already failed (Infants that met intubation criteria) and also is used electively for extubation when nCPAP extubation has previously failed or infants with Prolonged mechanical ventilation (more than 15 days) with high respiratory parameters (PMAP > 10 cmH2O and FiO2>35%).

DETAILED DESCRIPTION:
SNIPPV is used to prevent Intubation in Infants in which nCPAP has already failed (Infants that met intubation criteria) and also is used electively for extubation when nCPAP extubation has previously failed or infants with Prolonged mechanical ventilation (more than 15 days) with high respiratory parameters (PMAP > 10 cmH2O and FiO2>35%).

ELIGIBILITY:
Inclusion Criteria:

* Preterm Infants of less than 32 weeks of GA in which SNIPPV is applied for nCPAP failure.
* Preterm Infants of less than 32 weeks of GA in which SNIPPV is applied electively for extubation.

Exclusion Criteria: None

Ages: 1 Minute to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prospective observational study of SNIPPV use in preterm infants of less than 32 weeks of gestation from January 2012 to December of 2014.
  SNIPPV is used for:
  * nCPAP failure: Preterm infants supported with nCPAP that meet intubation criteria (FiO2>50%; apnea spells more than 4/h or more than 1 that needs PPV) if they are in a stable situation. SAP (systemic arterial pressure)> P10 with preserved respiratory drive (no more than 6 apneas episodes per hour or more than 2 requiring PPI).
  * Electively For extubation:
    * Preterm infants in which nCPAP extubation has previously failed or Prolonged mechanical ventilation (more than 15 days) with high respiratory parameters (PMAP > 10 cmH2O and FiO2>35%).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Avoid of Invasive Mechanical Ventilation in the next three days. | through study completion, an average of 1 year
  The rate of infants treated with non-invasisive ventilation that do not need to be intubated in the next three days.

SECONDARY OUTCOMES:
Time on MV | through study completion, an average of 1 year
  Days on MV during hospitalitation
Neurological impairment | through study completion, an average of 1 year
  Intraventricular hemorrhage grade 3 or 4 (papile´s classification)
Rate of patients with air leaks | through study completion, an average of 1 year
  pulmonary air leak

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramos-Navarro, Principal Investigator — Gregorio Marañón Hospital
Locations (1):
- Cristina Ramos-Navarro, Madrid, Spain